CLINICAL TRIAL: NCT05154253
Title: Augmenting Ankle Plantarflexor Function and Walking Capacity in Children With Cerebral Palsy
Brief Title: Augmenting Ankle Plantarflexor Function in Cerebral Palsy
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Northern Arizona University (Other)
Collaborators: Gillette Children's Specialty Healthcare (Other); University of Washington (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1R01HD107277 (NIH)
Record Dates: First submitted 2021-10-13; First posted 2021-12-13 (Actual); Last update posted 2024-02-28 (Actual); Status verified 2024-02

CONDITIONS: Cerebral Palsy
Keywords: Gait; Rehabilitation
MeSH Terms: conditions — Cerebral Palsy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (6):
- Device resisted gait training (treatment) (Experimental): We will conduct a randomized controlled trial (treatment vs. control) to compare functional outcomes following bilateral targeted ankle resistance training (2 visits/week for 12 weeks) vs. dose-matched standard functional gait training.
  Interventions: Device: Biomotum Spark: Robotic ankle resistance
- Standard gait training (control) (Experimental): We will conduct a randomized controlled trial (treatment vs. control) to compare functional outcomes following bilateral targeted ankle resistance training (2 visits/week for 12 weeks) vs. dose-matched standard functional gait training.
  Interventions: Other: Standard gait training
- Comparison to Standard PT (within subjects control) (Experimental): We will use a within-subject repeated measures design to compare both gait training groups to matched standard physical therapy.
  Interventions: Other: Standard physical therapy
- Device assisted ambulation (Experimental): We will compare task capacity and performance with adaptive ankle assistance vs. standard ankle foot orthoses and vs. shod (no ankle aid).
  Interventions: Device: Biomotum Spark: Robotic ankle assistance
- Passive brace assisted ambulation (Experimental): We will compare task capacity and performance with adaptive ankle assistance vs. standard ankle foot orthoses and vs. shod (no ankle aid).
  Interventions: Device: Ankle foot orthosis
- No ankle aid ambulation (Experimental): We will compare task capacity and performance with adaptive ankle assistance vs. standard ankle foot orthoses and vs. shod (no ankle aid).
  Interventions: Other: Standard walking

INTERVENTIONS:
Device: Biomotum Spark: Robotic ankle assistance — A lightweight assistive wearable ankle robotic device.
  Arms: Device assisted ambulation
Device: Biomotum Spark: Robotic ankle resistance — A lightweight resistive wearable ankle robotic device.
  Arms: Device resisted gait training (treatment)
Other: Standard gait training — Standard gait training without a device.
  Arms: Standard gait training (control)
Device: Ankle foot orthosis — Standard ankle foot orthosis
  Arms: Passive brace assisted ambulation
Other: Standard physical therapy — Physical therapy without a device.
  Arms: Comparison to Standard PT (within subjects control)
Other: Standard walking — Walking without a device
  Arms: No ankle aid ambulation

SUMMARY:
The first specific aim is to quantify improvement in ankle muscle function and functional mobility following targeted ankle resistance gait training in ambulatory children with cerebral palsy (CP). The primary hypothesis for the first aim is that targeted ankle resistance training will produce larger improvements in lower-extremity motor control, gait mechanics, and clinical measures of mobility assessed four- and twelve-weeks post intervention compared to standard physical therapy and standard gait training. The second specific aim is to determine the efficacy of adaptive ankle assistance to improve capacity and performance during sustained, high-intensity, and challenging tasks in ambulatory children with CP. The primary hypothesis for the second aim is that adaptive ankle assistance will result in significantly greater capacity and performance during the six-minute-walk-test and graded treadmill and stair stepping protocols compared to walking with ankle foot orthoses and walking with just shoes.

DETAILED DESCRIPTION:
A child's ability to walk effectively is essential to their physical health and general well-being. Unfortunately, many children with cerebral palsy (CP), the most common cause of pediatric physical disability, have difficulty walking and completing higher-intensity ambulatory tasks. This leads to children with CP engaging in levels of habitual physical activity that are well below guidelines and those of children without disabilities, which in turn contributes to many secondary conditions, including metabolic dysfunction and cardiovascular disease. There is broad clinical consensus that plantarflexor dysfunction is a primary contributor to slow, inefficient, and crouched walking patterns in CP; individuals with CP need more effective treatments and mobility aids for plantarflexor dysfunction. To meet this need, this proposal aims to evaluate a holistic strategy to address impaired mobility from plantarflexor dysfunction in CP using a lightweight, dual-mode (assistive or resistive) wearable robotic device. This strategy combines two complementary techniques: (1) targeted ankle resistance for neuromuscular gait training that provides precision therapy to elicit long-term improvements in ankle muscle function, and (2) adaptive ankle assistance to make walking easier during sustained, high-intensity, or challenging tasks.

Aim 1: Quantify improvement in ankle muscle function and functional mobility following targeted ankle resistance gait training in ambulatory children with CP Approach - Repeated Measures (RM) and randomized controlled trial: The investigators will compare functional outcomes following targeted ankle resistance training (2 visits/week for 12 weeks) vs. dose-matched standard physical therapy (RM) and vs. dose-matched standard treadmill training (randomized controlled trial). Primary Hypothesis: Targeted ankle resistance training will produce larger improvements in lower-extremity motor control, gait mechanics, and clinical measures of mobility assessed four- and twelve-weeks post intervention compared to the control conditions.

Aim 2: Determine the efficacy of adaptive ankle assistance to improve capacity and performance during sustained, high-intensity, and challenging tasks in ambulatory children with CP Approach - Repeated Measures: The investigators will compare task capacity and performance with adaptive ankle assistance vs. standard ankle foot orthoses and vs. shod (no ankle aid) during (a) 6-minute-walk-test, (b) extended-duration over-ground walking (sustained), (c) graded treadmill (high-intensity), and (d) stair-stepping (challenging) protocols. Task capacity and performance will be measured by duration, metabolic cost, speed, and stride length, as applicable. Primary Hypothesis: Adaptive ankle assistance will result in significantly greater capacity and performance compared to the control conditions.

ELIGIBILITY:
Inclusion Criteria:

* Ages between 8 and 21 years old, inclusive. Diagnosis of CP and a pathological gait pattern caused by ankle dysfunction.
* Able to understand and follow simple directions (based on parent report, if needed) and walk at least 30 feet with or without a walking aid (Gross Motor Function Classification System (GMFCS) Level I-III).
* At least 20° of passive plantar-flexion range of motion.

Exclusion Criteria:

* Concurrent treatment other than those assigned during the study.
* A condition other than CP that would affect safe participation.
* Surgical intervention within 6 months of participation.

Ages: 8 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 36 (Estimated)
Dates: Start 2023-02-01 (Actual); Primary Completion 2026-05-08 (Estimated); Study Completion 2026-09-25 (Estimated)

PRIMARY OUTCOMES:
Change in preferred walking speed | Immediately after the intervention
  Participant's preferred walking speed compared after to before the intervention
Change in preferred walking speed | 2 weeks after the intervention
  Participant's preferred walking speed compared after to before the intervention
Change in preferred walking speed | 12 weeks after the intervention
  Participant's preferred walking speed compared after to before the intervention
Change in similarity of plantarflexor muscle activity | Immediately after the intervention
  Similarity of the plantarflexor muscle activity profile across the gait cycle, measured using surface electromyography (the measurement tool) of the soleus muscle, to the average unimpaired electromyography muscle activity profile, as calculated via cross-correlation coefficient. A higher value indicates greater similarity.
Change in similarity of plantarflexor muscle activity | 2 weeks after the intervention
  Similarity of the plantarflexor muscle activity profile across the gait cycle, measured using surface electromyography (the measurement tool) of the soleus muscle, to the average unimpaired electromyography muscle activity profile, as calculated via cross-correlation coefficient. A higher value indicates greater similarity.
Change in similarity of plantarflexor muscle activity | 12 weeks after the intervention
  Similarity of the plantarflexor muscle activity profile across the gait cycle, measured using surface electromyography (the measurement tool) of the soleus muscle, to the average unimpaired electromyography muscle activity profile, as calculated via cross-correlation coefficient. A higher value indicates greater similarity.
Change in 6-minute-walk-test distance | Immediately after the intervention
  Distance traveled in 6 minutes during a 6-minute-walk-test protocol. A longer distance indicates greater walking capacity.
Change in 6-minute-walk-test distance | 2 weeks after the intervention
  Distance traveled in 6 minutes during a 6-minute-walk-test protocol. A longer distance indicates greater walking capacity.
Change in 6-minute-walk-test distance | 12 weeks after the intervention
  Distance traveled in 6 minutes during a 6-minute-walk-test protocol. A longer distance indicates greater walking capacity.
Change in variance in muscle activity | Immediately after the intervention
  Variance in muscle activity accounted for by one muscle synergy assessed using surface electromyography (the measurement tool) of the soleus, tibialis anterior, medial hamstrings, and vastus medialis. Muscle synergies will be computed from non-negative matrix factorization. Lower variance accounted for by one muscle synergy indicates a desired greater complexity of motor control.
Change in variance in muscle activity | 2 weeks after the intervention
  Variance in muscle activity accounted for by one muscle synergy assessed using surface electromyography (the measurement tool) of the soleus, tibialis anterior, medial hamstrings, and vastus medialis. Muscle synergies will be computed from non-negative matrix factorization. Lower variance accounted for by one muscle synergy indicates a desired greater complexity of motor control.
Change in variance in muscle activity | 12 weeks after the intervention
  Variance in muscle activity accounted for by one muscle synergy assessed using surface electromyography (the measurement tool) of the soleus, tibialis anterior, medial hamstrings, and vastus medialis. Muscle synergies will be computed from non-negative matrix factorization. Lower variance accounted for by one muscle synergy indicates a desired greater complexity of motor control.
Change in stride length | Immediately after the intervention
  Participant stride length during walking. Longer stride length is desired.
Change in stride length | 2 weeks after the intervention
  Participant stride length during walking. Longer stride length is desired.
Change in stride length | 12 weeks after the intervention
  Participant stride length during walking. Longer stride length is desired.
Change in stride-to-stride variability stride length | Immediately after the intervention
  Stride-to-stride variability of lower-extremity muscle activity for the soleus, tibias anterior, vastus lateralis, and medial hamstrings, measured via surface electromyography and calculated as the variance ratio across strides.
Change in stride-to-stride variability stride length | 2 weeks after the intervention
  Stride-to-stride variability of lower-extremity muscle activity for the soleus, tibias anterior, vastus lateralis, and medial hamstrings, measured via surface electromyography and calculated as the variance ratio across strides.
Change in stride-to-stride variability stride length | 12 weeks after the intervention
  Stride-to-stride variability of lower-extremity muscle activity for the soleus, tibias anterior, vastus lateralis, and medial hamstrings, measured via surface electromyography and calculated as the variance ratio across strides.
Change in walking posture | Immediately after the intervention
  Peak Lower-extremity joint angles summed across the ankle, knee, and hip joints, measured using motion capture (the measurement tool).
Change in walking posture | 2 weeks after the intervention
  Peak Lower-extremity joint angles summed across the ankle, knee, and hip joints, measured using motion capture (the measurement tool).
Change in walking posture | 12 weeks after the intervention
  Peak Lower-extremity joint angles summed across the ankle, knee, and hip joints, measured using motion capture (the measurement tool).
Change in Gross Motor Function Measure-66 sec. D&E | Immediately after the intervention
  Gross Motor Function Measure - 66, sections (D) standing, and (E) walking, running and jumping. Higher scores are better, and range from 0-3 for each measure.
Change in Gross Motor Function Measure-66 sec. D&E | 2 weeks after the intervention
  Gross Motor Function Measure - 66, sections (D) standing, and (E) walking, running and jumping. Higher scores are better, and range from 0-3 for each measure.
Change in Gross Motor Function Measure-66 sec. D&E | 12 weeks after the intervention
  Gross Motor Function Measure - 66, sections (D) standing, and (E) walking, running and jumping. Higher scores are better, and range from 0-3 for each measure.
Change in plantar-flexor strength | Immediately after the intervention
  Plantar-flexor muscle strength measured via hand-held dynamometry.
Change in plantar-flexor strength | 2 weeks after the intervention
  Plantar-flexor muscle strength measured via hand-held dynamometry.
Change in plantar-flexor strength | 12 weeks after the intervention
  Plantar-flexor muscle strength measured via hand-held dynamometry.
Distance traveled | 1 day
  Distance traveled during the 6-minute-walk-test, and treadmill and stair stepper bruce protocols.
Metabolic cost of transport from indirect calorimetry | 1 day
  Metabolic cost estimated from a wearable indirect calorimetry system during the 6-minute-walk-test, and treadmill and stair stepper bruce protocols
Subject perceived exertion | 1 day
  Subject perceived exertion (validated pictorial pediatric exertion scale). The scale is from 1-10, where a higher number indicates more effort.
Average muscle activity | 1 day
  Average stance-phase plantar flexor muscle activity assessed through surface electromyography of the soleus muscle.
Heart Rate | 1 day
  Average heart rate during each testing condition measured via chest-mounted heart rate monitor.

CONTACTS AND LOCATIONS:
Overall Officials: Zach F Lerner, PhD, Principal Investigator — Northern Arizona University
Locations (1):
- Gillette Children's Specialty Healthcare, Minneapolis, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Informed Consent Form (2023-03-06): https://cdn.clinicaltrials.gov/large-docs/53/NCT05154253/ICF_000.pdf